CLINICAL TRIAL: NCT04762563
Title: The Effect of Instrument Assisted Soft Tissue Mobilization and Kinesiology Taping on Connective Tissue Thickness in Patients With Chronic Low Back Pain
Brief Title: Effect of Treatment on Connective Tissue in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Medical Park Hospital Istanbul (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain; Connective Tissue Defect (Diagnosis)
MeSH Terms: conditions — Low Back Pain; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Study Group (Experimental): Patients in the IASTM group were asked to lie face down on a stretcher, exposing the entire lumbar region. IASTM was applied to all paraspinal muscles for a total of 5 minutes after massage cream was applied. Immediately afterwards, the same application was performed for the right and left hamstring muscles from the gluteal line to the bottom of the popliteal fossa for 3 minutes after massage cream was applied. IASTM application was performed vertically, horizontally and diagonally using instruments of different sizes and shapes at an angle of 45 degrees to the skin surface.
  Interventions: Other: IASTM application
- Active Comparator (Active Comparator): KT application (Kinesio Tape® Tex Gold) was performed using the "muscle technique". In lumbar region application, while the patient was standing, the tape was cut as a Y-strip with a base of 5 cm.
  Interventions: Other: Kinesio Tape® Tex Gold)

INTERVENTIONS:
Other: IASTM application — IASTM application .
  Arms: Experimental: Study Group
Other: Kinesio Tape® Tex Gold) — Kinesio Tape® Tex Gold)
  Arms: Active Comparator

SUMMARY:
The purpose of the study is to investigate the effects of instrument assisted soft tissue mobilization (IASTM) and kinesiology taping (KT) that are additional treatment to the conservative treatment for the lumbar region and hamstrings and connective tissue thickness in patients with chronic non-specific low back pain (CNSLBP).

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 30 and 50
* who had low back pain for at least 12 weeks,
* received no physical therapy in the last 6 months,
* received no IASTM or chemotherapy,
* had normal movement of the hip joint
* Visual Analog Scale value above 3

Exclusion Criteria:

* the presence of allergy and skin diseases,
* pregnancy,
* major structural spinal deformity (scoliosis, kyphosis, stenosis),
* inflammatory disease,
* presence of extruded and sequestered herniation, -signs of neurological disease, -
* presence of orthopedic diseases such as fracture
* a history of spinal surgery.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
straight leg test | 4 weeks
  Straight leg raise (SLR) was used to determine hamstring shortness. For SLR application, while the patient was lying on the back, the leg was lifted by the researcher to the level where the pain began, and the flexion angle in the hip was recorded
sit and reach test | 4 weeks
  The sit and reach test (SRT) to measure the flexibility.During SRT application, the distance between the middle fingers of the hands and the feet was recorded while the patient was in the long sitting position in the bed and reached the toes with their hands without bending the knees
Modified Schober test | 4 weeks
  Modified Schober Test and finger-ground distance evaluation for the spinal mobility assessment. For the Modified Schober Test, after marking 5 cm below and 10 cm above the spinous process of the lumbar vertebra while the patient was standing, the patient was asked to bend forward without bending the knees, and the change in the same range was recorded
finger-ground distance measurement | 4 weeks
  While measuring "finger-ground distance", the patient was asked to touch the ground with both hands while standing with the knees in extension. The distance between the fingertip and the ground was recorded
Ultrasonography | 4 weeks
  In this study, Siemens Acuson S 3000 device and Siemens HD 10 MHz linear probe were used for subcutaneous and perimuscular zone measurements.2 cm lateral to the midpoint of the L2-3 interspinous ligament is the area where the fascia planes are most parallel to the skin. In this study, the probe was centered at this point, which was determined while the patient was lying face down on the stretcher, and measurements were made from the right and left. For the measurement location in the hamstring region, the point where the fascia planes were most parallel to the skin was determined, as in the lumbar region. Measurement was performed in the area where the zones were most clearly seen lateral to the popliteal fossa.

CONTACTS AND LOCATIONS:
Locations (1):
- Emine Atıcı, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided